CLINICAL TRIAL: NCT03684785
Title: Merkel Cell Carcinoma, Cutaneous Squamous Cell Carcinoma, or Other Advanced Solid Tumors: A Phase 1b/2 Study of Cavrotolimod Combined With Pembrolizumab or Cemiplimab
Brief Title: Intratumoral Cavrotolimod Combined With Pembrolizumab or Cemiplimab in Patients With Merkel Cell Carcinoma, Cutaneous Squamous Cell Carcinoma, or Other Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was canceled for administrative reasons.
Sponsor: Exicure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AST-008-102
Record Dates: First submitted 2018-09-19; First posted 2018-09-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Advanced or Metastatic Merkel Cell Carcinoma; Advanced or Metastatic Cutaneous Squamous Cell Carcinoma; Advanced or Metastatic Melanoma; Advanced or Metastatic Head and Neck Squamous Cell Carcinoma; Advanced or Metastatic Solid Tumors
Keywords: Advanced or Metastatic Merkel Cell Carcinoma; Advanced or Metastatic Cutaneous Squamous Cell Carcinoma; Advanced or Metastatic Head and Neck Squamous Cell Carcinoma; Advanced or Metastatic Melanoma; Advanced or Metastatic Solid Tumors; Head and Neck; Squamous Cell Carinoma; Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Melanoma; Skin Cancer
MeSH Terms: conditions — Carcinoma, Merkel Cell; Melanoma; Skin Neoplasms | interventions — pembrolizumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation Phase 1b (Experimental): Determine the recommended Phase 2 dose of cavrotolimod in combination with pembrolizumab.
  Interventions: Drug: Cavrotolimod; Biological: Pembrolizumab
- Dose Expansion Phase 2; Merkel cell carcinoma (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and pembrolizumab in patients with advanced Merkel cell carcinoma that have progressed on an anti-PD-1 / anti-PD-L1 therapy.
  Interventions: Drug: Cavrotolimod; Biological: Pembrolizumab
- Dose Expansion Phase 2, cutaneous squamous cell carcinoma (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and cemiplimab in patients with advanced cutaneous squamous cell carcinoma that have progressed on an anti-PD-1.
  Interventions: Drug: Cavrotolimod; Biological: Cemiplimab
- Exploratory Phase 2, Merkel cell carinoma (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and pembrolizumab in patients with advanced Merkel cell carcinoma that have progressed on anti-PD-1 / anti-PD-L1 therapy.
  Interventions: Drug: Cavrotolimod; Biological: Pembrolizumab
- Exploratory Phase 2, Subcutaneous Dosing Cohort (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and pembrolizumab in patients with no cutaneous, subcutaneous, or accessible nodal tumor lesions amenable that have progressed on anti-PD-1 / anti-PD-L1 therapy.
  Interventions: Biological: Pembrolizumab; Drug: Cavrotolimod
- Exploratory Phase 2, Melanoma (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and pembrolizumab in patients with locally Advanced or Metastatic Melanoma that have progressed on anti-PD-1 / anti-PD-L1 therapy.
  Interventions: Drug: Cavrotolimod; Biological: Pembrolizumab
- Exploratory Phase 2, Liver Lesion (Experimental): Determine the safety and preliminary efficacy of cavrotolimod and pembrolizumab in patients with metastatic solid tumors with liver metastases that have progressed on anti-PD-1 / anti-PD-L1 therapy.
  Interventions: Drug: Cavrotolimod; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Cavrotolimod — Intratumorally dosed cavrotolimod.
  Arms: Dose Escalation Phase 1b; Dose Expansion Phase 2, cutaneous squamous cell carcinoma; Dose Expansion Phase 2; Merkel cell carcinoma; Exploratory Phase 2, Liver Lesion; Exploratory Phase 2, Melanoma; Exploratory Phase 2, Merkel cell carinoma
Biological: Pembrolizumab — Pembrolizumab dosing as per the US prescribing information.
  Arms: Dose Escalation Phase 1b; Dose Expansion Phase 2; Merkel cell carcinoma; Exploratory Phase 2, Liver Lesion; Exploratory Phase 2, Melanoma; Exploratory Phase 2, Merkel cell carinoma; Exploratory Phase 2, Subcutaneous Dosing Cohort
Biological: Cemiplimab — Cemiplimab dosing as per the US prescribing information.
  Arms: Dose Expansion Phase 2, cutaneous squamous cell carcinoma
Drug: Cavrotolimod — Subcutaneously dosed cavrotolimod
  Arms: Exploratory Phase 2, Subcutaneous Dosing Cohort

SUMMARY:
This is a phase 1b/2, open-label, two-part, multicenter trial designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of intratumoral cavrotolimod injections alone and in combination with intravenous pembrolizumab or cemiplimab in patients with Merkel Cell Carcinoma, cutaneous squamous cell carcinoma, and advanced solid tumors.

Phase 1b of this trial is a 3+3 dose escalation study evaluating escalating or intermediate dose levels of cavrotolimod given with a fixed dose of pembrolizumab.

The Phase 2 dose expansion part of the study will consist of two primary cohorts of patients: Merkel cell carcinoma and cutaneous squamous cell carcinoma. Patients in the Merkel Cell Carcinoma cohort will receive IT cavrotolimod combined with a fixed, standard dose of pembrolizumab while the Cutaneous Squamous Cell Carcinoma cohort will receive IT cavrotolimod combined with a fixed, standard dose of cemiplimab. The Phase 2 dose expansion is designed to provide a preliminary estimate of efficacy in patients that have progressed on an anti-PD-(L)1 CPI.

DETAILED DESCRIPTION:
This study will be conducted in 2 phases. Phase 1 evaluates cavrotolimod given in combination with pembrolizumab in patients with advanced solid tumors in a classical 3+3 dose escalation design, with up to five ascending dose cohorts of cavrotolimod and enrollment of at least 3 patients per cohort to identify an RP2D. Patients will be dosed twice with cavrotolimod as a monotherapy before adding pembrolizumab, which will be added starting at the second cycle. Once the MTD or highest escalation cohort has been reached, or notable efficacy has been observed at a given dose level, and a decision as to a RP2D has been made, a two 2-stage expansion cohort design will be initiated.

Phase 2 will evaluate the RP2D of cavrotolimod given in combination with pembrolizumab or cemiplimab in two expansion cohorts following a modified Simon 2-stage optimal design comprised of patients with Merkel cell carcinoma or cutaneous squamous cell carcinoma. who previously received and have progressed on an anti-PD-(L)1 CPI. Patients in the Merkel Cell Carcinoma cohort will receive IT cavrotolimod combined with a fixed, standard dose of pembrolizumab while the Cutaneous Squamous Cell Carcinoma cohort will receive IT cavrotolimod combined with a fixed, standard dose of cemiplimab.

Phase 2 will include an exploratory expansion cohort to evaluate cavrotolimod in combination with pembrolizumab in patients with other advanced solid tumors, including melanoma, who have progressed on anti-PD-(L)1 therapy.

Exploratory expansion cohorts will evaluate patients with melanoma and additional patients with Merkel Cell Carcinoma who do not meet criteria for enrollment in the primary Merkel Cell Carcinoma cohort. In addition, two exploratory cohorts have been added to evaluate patients with advanced solid tumors and no superficial tumor accessible for IT injection using subcutaneously administered cavrotolimod or IT injection into liver metastases.

A cohort of up to 10 evaluable patients with locally advanced or metastatic solid tumors with no cutaneous, subcutaneous, or accessible nodal tumor lesions available for IT injection may be enrolled (inclusion criterion #4). The inclusion/exclusion criteria for this exploratory cohort will otherwise be the same as those used for the Phase 2 dose expansion cohorts except these patients will not be required to have a lesion accessible for biopsy (inclusion criterion #5). Patients will be dosed with cavrotolimod subcutaneously at a dose not to exceed the recommended Phase 2 dose, 32 mg, in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female ≥18 years of age.
3. Must have an advanced inoperable histologically diagnosed solid tumor.

   * Phase 2 Merkel Cell Carcinoma Dose Expansion Cohort: locally advanced or metastatic Merkel cell caricinoma
   * Phase 2 Cutaneous Squamous Cell Carcinoma Dose Expansion Cohort: locally advanced or metastatic cutaneous squamous cell carcinoma
   * Phase 2 Merkel Cell Carcinoma Exploratory Expansion Cohort: locally advanced or metastatic Merkel cell carcinoma
   * Phase 2 Melanoma Exploratory Expansion Cohort: Locally advanced or metastatic melanoma
   * Phase 2 Subcutaneous Dosing Exploratory Cohort: Locally advanced or metastatic solid tumors
   * Phase 2 Liver Lesion Exploratory Cohort: metastatic solid tumors with liver metastases
4. Phase 1b, Phase 2 Merkel Cell Carcinoma Dose Expansion Cohort, Phase 2 Cutaneous Squamous Cell Carcinoma Dose Expansion Cohort, Phase 2 Merkel Cell Carcinoma Exploratory Expansion Cohort, Phase 2 Melanoma Exploratory Expansion Cohort:

   At least one tumor lesion amenable to repeated IT injection via palpation or ultrasound. Injection of deep visceral lesions is not permitted.

   Patients enrolled in subcutaneous dosing cohort do not need lesions amenable to subcutaneous dosing.
5. Phase 1b and Phase 2 Melanoma Exploratory Expansion Cohort:

   Agrees to provide a newly obtained biopsy of one or two lesions, and agrees to repeat biopsies, if applicable.
6. Phase 1b:

   In the investigator's opinion the patient may derive clinical benefit from the treatment or is ineligible for a particular form of standard therapy due to tolerability, or the patient failed one or more established standard medical anti-cancer therapies. Exposure to anti-PD-(L)1 or anti-CTLA-4 antibody CPIs is permitted but not required.

   Phase 2 Merkel Cell Carcinoma Dose Expansion Cohort:

   i. At least a minimum number of cycles of avelumab, nivolumab, or pembrolizumab. Prior anti-CTLA-4 antibody therapy, including as most recent preceding therapy in combination with avelumab or pembrolizumab, is permitted but not required.

   ii. Confirmed progressive disease during treatment with avelumab or pembrolizumab therapy,

   Phase 2 Cutaneous Squamous Cell Carcinoma Dose Expansion Cohort

   i. At least a minimum number of cycles of cemiplimab, nivolumab, or pembrolizumab. Prior ipilimumab therapy, including as most recent preceding therapy in combination with cemiplimab, nivolumab, or pembrolizumab, is permitted but not required.

   ii. Confirmed progressive disease on cemiplimab or pembrolizumab therapy

   Phase 2 MCC and Melanoma Exploratory Expansion Cohort and Phase 2 Subcutaneous Dosing Exploratory Expansion Cohort:

   i. Treatment duration with anti-PD-(L)1 antibody ≥8 weeks as the most recent preceding therapy prior to being enrolled in this study with confirmed progression. Anti-PD-(L)1 was administrated for metastatic or locally advanced Merkel Cell Carcinoma or melanoma. Prior ipilimumab therapy, including as most recent therapy in combination with anti-PD-(L)1 therapy, is permitted but not required.

   ii. Confirmed progressive disease on anti-PD-(L)1 antibody therapy
7. Phase 1b and Phase 2 Melanoma Exploratory Expansion Cohort:

   Evaluable disease per RECIST 1.1 with at least two target lesions as defined by RECIST 1.1. Both injectable and non-injectable target lesions should be chosen for efficacy evaluation.
8. For the Phase 2 expansion portions of the study, a maximum of 4 prior lines of systemic treatment for locally advanced or metastatic disease.

   * Phase 2 Merkel Cell Carcinoma and Melanoma Exploratory Expansion Cohorts and Phase 2 Subcutaneous Dosing Exploratory Cohort
9. For female patients of childbearing potential, defined as females who 1) have not undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy or 2) have not been postmenopausal for at least 12 consecutive months [i.e., have had menses at any time during the preceding 12 consecutive months]):

   • Willing to use one of the following effective methods of contraception for at least 30 days before administration of cavrotolimod, during treatment with cavrotolimod, pembrolizumab, or cemiplimab, and for at least four months after the last dose of cavrotolimod, pembrolizumab, or cemiplimab:

   i. Total abstinence from sexual intercourse with a partner that may result in pregnancy

   ii. Hormonal contraception (oral, parenteral, or transdermal) used for at least 3 consecutive months prior to the first dose of cavrotolimod

   iii. Intrauterine contraceptive device

   iiii. Barrier contraception (i.e., condom, cap, diaphragm, or sponge with spermicide)

   For male patients who have not had a vasectomy:

   • Willing to use one of the following effective methods of contraception for at least 30 days before administration of cavrotolimod, during treatment with cavrotolimod, pembrolizumab, or cemiplimab, and for at least four months after the last dose of cavrotolimod, pembrolizumab, or cemiplimab:

   i. Total abstinence from sexual intercourse with a female partner of childbearing potential

   ii. Use by female partner of hormonal contraception (oral, parenteral, or transdermal) for at least 3 consecutive months prior to the first dose of cavrotolimod

   iii. Use by female partner of intrauterine contraceptive device

   iiii. Barrier contraception (i.e., condom, cap, diaphragm, or sponge with spermicide)
10. Regarding history of CPI-related adverse events:

    i. Resolution of CPI-related AEs (including irAEs) to G0-1 and no corticosteroids for the amelioration of those irAEs for at least 4 weeks prior to the first dose of cavrotolimod. Controlled hypothyroidism and controlled adrenal insufficiency are exceptions to this criterion, provided doses do not exceed the threshold described in exclusion criterion #13.

    ii. No history of CTCAE G4 irAEs from CPI. iii. No history of CTCAE G3 irAEs from CPI. Patients with a history of CTCAE G3 irAEs from CPI requiring steroid treatment for no greater than 12 weeks may be considered at the discretion of the Investigator if supported by an assessment of risk-benefit and after discussion with the Medical Monitor.
11. Adequate organ function.
12. Able and willing to comply with the protocol and the restrictions and assessments therein.

Exclusion Criteria:

1. Small molecule or tyrosine kinase inhibitor within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of cavrotolimod, chemotherapy or biological cancer therapy within 3 weeks prior to the first dose of cavrotolimod, nitrosourea, or radioisotope within 6 weeks prior to first dose of cavrotolimod, or non-recovery to CTCAE G1 or better from the AEs due to cancer therapeutics administered more than 4 weeks earlier.
2. Known hypersensitivity to any phosphorothioate oligonucleotide, or previous exposure to a TLR9 agonist drug.
3. Previous severe hypersensitivity reaction to treatment with pembrolizumab, cemiplimab or another anti-PD-(L)1 monoclonal antibody.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) >1.
5. Symptomatic ascites or pleural effusion. A patient with these conditions who has received treatment such as therapeutic thoracentesis or paracentesis and is clinically stable, defined as not requiring repeat drainage procedure within 2 weeks, may be considered after discussion with the Medical Monitor.
6. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to the first dose of cavrotolimod, have no evidence of new or enlarging brain metastases and are off steroids for at least 14 days prior to the first dose of cavrotolimod.
7. Known history of a hematologic malignancy, malignant primary brain tumor or malignant sarcoma, or of another malignant primary solid tumor (other than that under study), with the following exceptions: 1) patients who have undergone potentially curative therapy with no evidence of that disease for 3 years prior to the first dose of cavrotolimod; 2) patients who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers; 3) stable chronic lymphocytic leukemia not requiring treatment within 3 years prior to the first dose of cavrotolimod.
8. Significant autoimmune disease that requires or required systemic steroids or immunosuppressive agents within the last year. The following are not exclusionary: 1) vitiligo, resolved asthma/atopy, and limited eczema; 2) conidtions requiring intermittent use of bronchodilators or local steroid injections; 3) hypothyroidism or adrenal insufficiency that is stable on hormone replacement; or 4) irAEs related to checkpoint inhibitor therapy, provided inclusion criterion #10 and exclusion criterion #11 are met.
9. Use of systemic corticosteroids to treat inflammatory or autoimmune symptoms within 15 days or other immunosuppressive drugs within 30 days prior to the first dose of cavrotolimod. Inhaled and topical corticosteroids are permitted. Up to 10 mg/day prednisone or equivalent is permitted for hypothyroidism or adrenal insufficiency.
10. Received an investigational product or been treated with an investigational device within 30 days prior to the first dose of cavrotolimod or will start any other investigational product or device study within 30 days after last study drug administration.
11. History or clinical evidence of any surgical or medical condition which the Investigator judges as likely to interfere with the results of the study or pose an additional risk in participating e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
12. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study through 4 months after the last dose of cavrotolimod, pembrolizumab, or cemiplimab.
13. Allergy or intolerance preventing use of H1 blockers (e.g., diphenhydramine, cetirizine) and H2 blockers (e.g., famotidine) used as antihistamine premedication prior to cavrotolimod injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Adverse events of cavrotolimod alone and in combination with pembrolizumab or cemiplimab | Study day 36
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Recommended Phase 2 dose | 12 months
  To recommend a dose of cavrotolimod and combination regimen for further development
Objective response rate (ORR) per RECIST v1.1 | 24 months
  ORR to be calculated overall and by cohort/subgroup using RECIST v1.1. Subgroups will be defined for the efficacy analyses based on prior exposure and response to immune checkpoint inhibitors.
Measure changes in correlative biomarkers including tumor-infiltrating lymphocytes, PD-L1 and other checkpoint expression at baseline, after cavrotolimod monotherapy, and after combination therapy of both cavrotolimod and pembrolizumab or cemiplimab. | Study day 36
  IHC on FFPE biopsies will be used to assess markers.
Measure changes in gene expression profiles at baseline, after cavrotolimod monotherapy, and after combination therapy of both cavrotolimod and pembrolizumab or cemiplimab. | Study day 36
  Selected gene-expression profiling on gene expression will be performed with nCounter (NanoString Technologies).

CONTACTS AND LOCATIONS:
Overall Officials: Exicure Inc., Study Director — Exicure, Inc.
Locations (26):
- United States (26):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California Irvine, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - John Wayne Cancer Institute / Providence St. John's Health Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Western States Cancer Center, Englewood, Colorado
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Cancer Center, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Valley - Mount Sinai Comprehensive Cancer Center, Paramus, New Jersey
  - Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center / Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sammons Cancer Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington- Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia Cancer Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices) will be shared to researchers who provide a methodologically sound proposal and sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Access will be considered to researchers who provide a methodologically sound proposal. Analysis must achieve the aims outlined in the approved proposal. Proposals should be directed to edegoma@exicuretx.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 36 months following article publication.

REFERENCES:
- [Derived] Milhem MM, Wise-Draper TM, Chandra S, Hanna GJ, Laux DE, Medina TM, Ansstas G, Daud A, Kelly CM, O'Day SJ, Perez CA, Wong MK, Friedlander PA, Kristedja TS, Burgess MA, Cowey CL, Hanks BA, Weight RM, Daniel WL, Feltner DE, Mix S, Sindelar L, Bexon AS, Bexon MF, Michel RE, Bhatia S. Phase 1b/2 study evaluating safety, efficacy and immune effects of TLR9 agonist cavrotolimod with anti-PD-1 antibodies among patients with advanced solid tumors. J Immunother Cancer. 2025 Jul 25;13(7):e011651. doi: 10.1136/jitc-2025-011651. PMID 40713179
- See also: Exicure homepage — http://www.exicuretx.com